CLINICAL TRIAL: NCT02625857
Title: An Open-Label, Phase 1 Study of the Safety and Immunogenicity of JNJ-64041809, a Live Attenuated Listeria Monocytogenes Immunotherapy, in Subjects With Metastatic Castration-resistant Prostate Cancer
Brief Title: Safety & Immunogenicity of JNJ-64041809, a Live Attenuated Double-deleted Listeria Immunotherapy, in Participants With Metastatic Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107668; 64041809PCR1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: Prostatic Neoplasms, Castration-Resistant; JNJ-64041809; Listeria monocytogenes
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Cohort 1A and 1B (Experimental): JNJ-64041809 will be administered intravenously (IV) once every 21 days.
  Interventions: Biological: JNJ-64041809 (Cohort 1A and 1B)
- Dose Cohort 2A and 2B (Experimental): JNJ-64041809 will be administered intravenously (IV) once every 21 days.
  Interventions: Biological: JNJ-64041809 (Cohort 2A and 2B)

INTERVENTIONS:
Biological: JNJ-64041809 (Cohort 1A and 1B) — JNJ-64041809 will be administered IV at a lower dose in Cohort 1A (1x10^8 colony forming units [CFU]) and at a higher dose in Cohort 1B (1x10^9 CFU).
  Arms: Dose Cohort 1A and 1B
Biological: JNJ-64041809 (Cohort 2A and 2B) — JNJ-64041809 will be administered intravenously (IV) once every 21 days at the recommended dose as determined in Cohort 1A or 1B.
  Arms: Dose Cohort 2A and 2B

SUMMARY:
The purpose of this study is to find and evaluate the recommended Phase 2 dose (RP2D) of JNJ-64041809, a live attenuated double deleted (LADD) Listeria monocytogenes (bacteria in which two virulence genes, which encode molecules that help cause disease, have been removed) when administered intravenously to participants with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1, open-label, multicenter and 2-part study. The Part 1 of study will be Dose Escalation phase to determine the recommended Phase 2 dose (RP2D) based on safety and pharmacodynamic assessments and Part 2 will be Dose Expansion Phase to evaluate 2 expansion cohorts (Cohort 2A and 2B) after the RP2D for JNJ-64041809 is determined in Part 1. The study will consist of a Screening Period (from signing of informed consent until immediately before the first dose), an open-label Treatment Period (from the first dose of study drug until the End-of-Treatment Visit); and a Post treatment Follow-up Period (after the End-of Treatment Visit until study discontinuation). Participants will be primarily evaluated for RP2D. Participants safety will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate with progressive metastatic disease which, in the opinion of the investigator, requires initiation of new treatment. The assessment of disease progression can be based on either PSA rise, new or progressive soft tissue disease (based on computed tomography [CT] or magnetic resonance imaging [MRI] scans), or new or progressive bony disease based on radionuclide bone scan or 18F-sodium fluoride positron emission tomography/computed tomography [NaF PET/CT] scans). Participants being considered for Cohort 2B must, in addition, have primary or metastatic lesions amenable to tumor biopsies
* Must have received at least 2 prior approved therapies
* Ongoing androgen depletion therapy with a Gonadotropin Releasing Hormone analog or inhibitor, or orchiectomy (surgical or medical castration)
* Serum testosterone levels less than (<) 50 nanogram per deciliter (ng/dL) determined within 4 weeks prior to start of study drug
* For participants previously treated with first generation anti-androgens (ie, flutamide, nilutamide, or bicalutamide), discontinuation of flutamide or nilutamide therapy must occur greater than (>) 4 weeks (>6 weeks for bicalutamide) prior to start of study drug with no evidence of an anti-androgen withdrawal response (no decline in serum PSA)

Exclusion Criteria:

* Untreated brain metastases. Participants must have completed treatment for brain metastasis, and be neurologically stable off steroids, for at least 28 days prior to first dose of study drug
* Untreated spinal cord compression
* History of listeriosis or vaccination with a listeria-based vaccine or prophylactic vaccine (example influenza, pneumococcal, diphtheria, tetanus, and pertussis [dTP/dTAP]) within 28 days of study treatment
* Known allergy to both penicillin and trimethoprim/sulfamethoxazole. Participants who are allergic to only one of these antibiotics are allowed to enroll
* Concurrent treatment with anti -Tumor necrosis factor (TNF) alpha therapies, systemic corticosteroids (prednisone dose >10 mg per day or equivalent) or other immune suppressive drugs within the 2 weeks prior to Screening. Steroids that are topical, inhaled, nasal (spray), or ophthalmic solution are permitted

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence of Dose-limiting-toxicity (DLT) | first 21 days after the first infusion
  Percentage of Participants who Experienced DLT will be evaluated. The DLT dose level is defined as an unacceptable level of toxicity as evidenced by a DLT rate of greater than or equal to (>=) 33 percent (%).
Part 2: Antigen-specific T-cell Response | up to 1 year
  Biomarker studies will be performed to evaluate immune responses to the vaccine after the first intravenous (IV) immunization.
Part 1 and Part 2: Incidence of Adverse Events (AEs) | From signing of informed consent form to 30 days after last dose of study drug
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Incidence was defined as the number of participants who experienced an adverse event within their period of participation in this study. Incidence of adverse events will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).

SECONDARY OUTCOMES:
Part 1 and Part 2: Objective Response Rate (ORR) | Baseline up to 30 days after last dose of study drug
  Objective response rate is defined as the percentage of participants who achieve complete response (CR) or partial response (PR), as assessed by the investigator.
Part 1 and Part 2: Duration of Response (DOR) | Baseline up to 30 days after last dose of study drug
  Duration of response will be calculated from the date of initial documentation of a response (CR or PR) to the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death.
Part 1 and Part 2: Progression-free Survival (PFS) | Baseline up to 30 days after last dose of study drug
  Progression-free survival is defined as the duration from the date of first dose of study drug until the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death, whichever comes first.
Part 1 and Part 2: Time to Prostate Specific Antigen (PSA) progression (TTPP) | Baseline up to 30 days after last dose of study drug
  Time to PSA progression is measured from the date of first dose of study drug until the date of PSA progression according to the Prostate Cancer Clinical Trials Working Group (PCWG2) criteria.
Part 1 and Part 2: Blood Culture Assessment of JNJ-64041809 | Periodically during treatment and up to one year after End of Treatment (EOT) visit
  This assessment will include the reporting of surveillance blood cultures (peripherally drawn, and through venous access device [if applicable]) for 1 year after the completion of JNJ-64041809 therapy.
Part 1 and Part 2: Shedding Profile of JNJ-64041809 From Cultured Samples of Feces, Urine, and Saliva | During cycle 1 (up to 21 days of treatment period) and at EOT visit (within 30 days after last dose)
  The shedding of JNJ-64041809 will be studied in cultures of (1) feces by stool or rectal swab, (2) urine samples, and (3) saliva samples.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- United States (6):
  - San Francisco, California
  - Baltimore, Maryland
  - St Louis, Missouri
  - Nashville, Tennessee
  - Houston, Texas
  - Madison, Wisconsin

REFERENCES:
- [Background] Le DT, Dubenksy TW Jr, Brockstedt DG. Clinical development of Listeria monocytogenes-based immunotherapies. Semin Oncol. 2012 Jun;39(3):311-22. doi: 10.1053/j.seminoncol.2012.02.008. PMID 22595054
- [Background] Brockstedt DG, Giedlin MA, Leong ML, Bahjat KS, Gao Y, Luckett W, Liu W, Cook DN, Portnoy DA, Dubensky TW Jr. Listeria-based cancer vaccines that segregate immunogenicity from toxicity. Proc Natl Acad Sci U S A. 2004 Sep 21;101(38):13832-7. doi: 10.1073/pnas.0406035101. Epub 2004 Sep 13. PMID 15365184